CLINICAL TRIAL: NCT01503333
Title: Girls on the Move Intervention
Brief Title: Girls on the Move Intervention to Increase Physical Activity Among Middle School Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Lorraine Robbins, Associate Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HL109101 (NIH)
Record Dates: First submitted 2011-12-23; First posted 2012-01-04 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Physical Activity
Keywords: exercise; adolescent; intervention; female; counseling
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): The control condition will complete data collection activities and receive their usual school offerings.
- Physical activity intervention (Experimental): Receiving Physical activity intervention which includes individual counseling with the school nurse, tailored feedback from computer program, and after-school physical activity club.
  Interventions: Behavioral: Physical activity intervention

INTERVENTIONS:
Behavioral: Physical activity intervention — Receiving individual counseling with the school nurse, tailored feedback from computer program, and after-school physical activity club.
  Arms: Physical activity intervention

SUMMARY:
The purpose of this school-based trial is to test the efficacy of an intervention to increase moderate to vigorous physical activity (MVPA) among middle school girls. The 17-week "Girls on the Move" (GOTM) intervention has 3 components. Two individual-level components occurring during school hours include: (1) two face-to-face motivational, individually tailored counseling sessions with a school nurse, and (2) an interactive Internet-based session during which each girl receives motivational, individually tailored feedback messages (at 9 weeks). A group-level component, 90-minute Physical Activity (PA) Club provides an important venue after school that includes activities to assist girls in establishing a behavioral pattern of MVPA. The control condition will complete data collection activities and receive their usual school offerings.

The investigators hypothesize that immediately post-intervention, minutes of MVPA will be greater by 16 min./wk. in the intervention than control group; At 9 months post-intervention follow-up, minutes of MVPA will be greater in the intervention than control group; and immediately post-intervention, cardiovascular (CV) fitness will be higher and body mass index (BMI) and percent body fat will be lower in the intervention than control group.

DETAILED DESCRIPTION:
Our 17-week "Girls on the Move" (GOTM) intervention for middle school girls applies the Health Promotion Model (HPM) and Self-Determination Theory (SDT) and has 3 components. Two individual-level components occurring during school hours include: (1) two face-to-face motivational, individually tailored counseling sessions with a school nurse (occurring at baseline and near 17 wks.), and (2) an interactive Internet-based session during which each girl receives motivational, individually tailored feedback messages (at 9 wks.). A group-level component, 90-min. PA Club, led by PA instructors (e.g., individuals from community; teachers, including physical education (PE); and sports team coaches) provides an important venue after school that includes MVPAs (requested by girls in pilot) to assist girls in establishing a behavioral pattern of MVPA. The control condition will complete data collection activities and receive their usual school offerings.

The purpose of this school-based group randomized trial (GRT) is to evaluate the efficacy of the comprehensive GOTM intervention to increase middle school girls' min. of MVPA and improve cardiovascular (CV) fitness, body mass index (BMI), and percent body fat (% BF) immediately post-intervention (after 17 wks.) and MVPA at 9-mo. follow-up (F/U; 9 mos. after end of intervention). Secondary analyses will examine if MVPA is mediated by cognitive (e.g., perceived benefits of PA, barriers to PA, and PA self-efficacy; social support) and affective variables (e.g., enjoyment of and motivation for PA).

Based on demographics of the urban schools, we expect a low-SES, mixed-race, predominately African American, sample. Eight schools will be randomly assigned to the PA intervention (n = 4) or comparison condition (n = 4) in the fall of yrs. 2, 3, and 4 (total N = 8 X 3 = 24 different schools). Sixty-two girls meeting inclusion criteria based on answers to a screening tool will be recruited in each school during each of the three yrs.

The long-term goal is to increase MVPA as a means to address the high overweight and obesity prevalence among adolescent girls.

ELIGIBILITY:
Inclusion Criteria:

* 5th- 6th- and 7th-grade girls (ages 9-14; 8th-graders if needed in middle schools having only 7th- and 8th- grades)
* Available and willing to participate in PA Club 3 days/wk. for 17wks.
* Available for follow-up (9 mos. after intervention ends)
* Agree to random assignment
* Able to read, understand, and speak English.

Exclusion Criteria:

* Involved in or planning to be involved in school or community sports or other organized PAs, such as dance lessons, that involve MVPA and require participation 3 or more days/wk. after school during every season of the school year
* A health condition precluding safe MVPA.

Ages: 9 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1543 (Actual)
Dates: Start 2011-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine B Robbins, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

REFERENCES:
- [Background] Robbins LB, Pfeiffer KA, Vermeesch A, Resnicow K, You Z, An L, Wesolek SM. "Girls on the Move" intervention protocol for increasing physical activity among low-active underserved urban girls: a group randomized trial. BMC Public Health. 2013 May 15;13:474. doi: 10.1186/1471-2458-13-474. PMID 23672272
- [Background] Ling J, Robbins LB, Resnicow K, Bakhoya M. Social support and peer norms scales for physical activity in adolescents. Am J Health Behav. 2014 Nov;38(6):881-9. doi: 10.5993/AJHB.38.6.10. PMID 25207514
- [Background] Vermeesch AL, Ling J, Voskuil VR, Bakhoya M, Wesolek SM, Bourne KA, Pfeiffer KA, Robbins LB. Biological and Sociocultural Differences in Perceived Barriers to Physical Activity Among Fifth- to Seventh-Grade Urban Girls. Nurs Res. 2015 Sep-Oct;64(5):342-50. doi: 10.1097/NNR.0000000000000113. PMID 26325276
- [Background] Robbins LB, Ling J, Wesolek SM, Kazanis AS, Bourne KA, Resnicow K. Reliability and Validity of the Commitment to Physical Activity Scale for Adolescents. Am J Health Promot. 2017 Jul;31(4):343-352. doi: 10.4278/ajhp.150114-QUAN-665. Epub 2016 Nov 17. PMID 26730556
- [Background] Gammon C, Pfeiffer KA, Kazanis A, Ling J, Robbins LB. Cardiorespiratory fitness in urban adolescent girls: associations with race and pubertal status. J Sports Sci. 2017 Jan;35(1):29-34. doi: 10.1080/02640414.2016.1154594. Epub 2016 Mar 4. PMID 26942487
- [Background] Robbins LB, Ling J, Toruner EK, Bourne KA, Pfeiffer KA. Examining reach, dose, and fidelity of the "Girls on the Move" after-school physical activity club: a process evaluation. BMC Public Health. 2016 Jul 30;16:671. doi: 10.1186/s12889-016-3329-x. PMID 27473613
- [Background] Bakhoya M, Ling J, Pfeiffer KA, Robbins LB. Evaluating Mailed Motivational, Individually Tailored Postcard Boosters for Promoting Girls' Postintervention Moderate-to-Vigorous Physical Activity. Nurs Res. 2016 Sep-Oct;65(5):415-20. doi: 10.1097/NNR.0000000000000173. PMID 27579509
- [Background] Ling J, Robbins LB. Psychometric Evaluation of Three Psychosocial Measures Associated With Physical Activity Among Adolescent Girls. J Sch Nurs. 2017 Oct;33(5):344-354. doi: 10.1177/1059840516685857. Epub 2016 Dec 29. PMID 28030983
- [Background] Voskuil VR, Pierce SJ, Robbins LB. Comparing the Psychometric Properties of Two Physical Activity Self-Efficacy Instruments in Urban, Adolescent Girls: Validity, Measurement Invariance, and Reliability. Front Psychol. 2017 Aug 3;8:1301. doi: 10.3389/fpsyg.2017.01301. eCollection 2017. PMID 28824487
- [Background] Robbins LB, Ling J, Resnicow K. Demographic differences in and correlates of perceived body image discrepancy among urban adolescent girls: a cross-sectional study. BMC Pediatr. 2017 Dec 6;17(1):201. doi: 10.1186/s12887-017-0952-3. PMID 29207976
- [Background] Robbins LB, Ling J, Dalimonte-Merckling DM, Sharma DB, Bakhoya M, Pfeiffer KA. Sources and Types of Social Support for Physical Activity Perceived by Fifth to Eighth Grade Girls. J Nurs Scholarsh. 2018 Mar;50(2):172-180. doi: 10.1111/jnu.12369. Epub 2017 Dec 21. PMID 29266689
- [Derived] Robbins LB, Ling J, Wen F. Moderators in a physical activity intervention for adolescent girls. Pediatr Res. 2020 Nov;88(5):810-817. doi: 10.1038/s41390-020-0818-5. Epub 2020 Mar 2. PMID 32120378
- [Derived] Pfeiffer KA, Robbins LB, Ling J, Sharma DB, Dalimonte-Merckling DM, Voskuil VR, Kaciroti N, Resnicow K. Effects of the Girls on the Move randomized trial on adiposity and aerobic performance (secondary outcomes) in low-income adolescent girls. Pediatr Obes. 2019 Nov;14(11):e12559. doi: 10.1111/ijpo.12559. Epub 2019 Jul 3. PMID 31267695
- [Derived] Robbins LB, Ling J, Sharma DB, Dalimonte-Merckling DM, Voskuil VR, Resnicow K, Kaciroti N, Pfeiffer KA. Intervention Effects of "Girls on the Move" on Increasing Physical Activity: A Group Randomized Trial. Ann Behav Med. 2019 Mar 28;53(5):493-500. doi: 10.1093/abm/kay054. PMID 29985968

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: The control condition completed data collection activities and received their usual school offerings, such as physical education.
- Physical Activity Intervention: The intervention group completed data collection activities and received the 17-week intervention which included 3 components to help the girls increase their physical activity: 1) two face-to-face motivational interviewing sessions (one at the beginning and the other near the end of the intervention period) with a school nurse/trained counselor; 2) motivational feedback tailored based on each girl's survey responses and delivered via an iPad shortly after the intervention midpoint; and 3) after-school physical activity club for 90 minutes 3 days per week at each girl's school.
  Physical activity intervention: Receiving individual counseling with the school nurse, tailored feedback from computer program, and after-school physical activity club.
Period: Overall Study
Arm/Group | Control | Physical Activity Intervention
Started | 777 | 766
Completed Baseline | 766 | 753
Completed Post-intervention | 680 | 706
Completed (Completed 9-month post-intervention follow-up measures) | 437 | 461
Not Completed | 340 | 305

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Physical Activity Intervention | Total
Number analyzed (Participants) | 766 | 753 | 1519
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 766 | 753 | 1519
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Single item multiple choice: How old are you? Population: 766 are in control group, and 753 are in intervention group.
  years | 12.05 (1.02) | 12.05 (0.99) | 12.05 (1.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 766 | 753 | 1519
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 90 | 111 | 201
  Not Hispanic or Latino | 629 | 603 | 1232
  Unknown or Not Reported | 47 | 39 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 6 | 13
  Asian | 15 | 26 | 41
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 416 | 340 | 756
  White | 198 | 214 | 412
  More than one race | 94 | 96 | 190
  Unknown or Not Reported | 34 | 71 | 105

OUTCOME MEASURES:

1. Primary Outcome: Minutes of Moderate to Vigorous Physical Activity (MVPA) Post-intervention
Description: Minutes of MVPA were measured via ActiGraph GT3X+ accelerometers worn on an elastic belt at the right hip for 7 consecutive days, including 5 weekdays and 2 weekend days at post-intervention. Monitors were set to start collecting and storing data in raw format beginning 5:00 A.M. on the day after they were distributed to girls each school. Data were re-integrated to 15-second epochs and processed using established intensity cut-points. One week after distribution, data collectors returned to each school to collect the accelerometers. The majority (1386 [post-intervention] of 1519 girls [baseline], 91.24%) provided at least 8 hours of data on 3 weekdays and 1 weekend day. An imputation approach based on all available data in hour blocks on all 7 days was implemented. Wear time was standardized to 14 hours/weekday (one hour before each school's actual start time; 7 hours during school; 6 hours after school) and 10 hours/weekend day (later awake time from 11 a.m. to 9 p.m.).
Time Frame: Minutes of moderate to vigorous physical activity per hour at post-intervention (after 17-week intervention)
Population: The majority (1386 [post-intervention] of 1519 girls [baseline], 91.24%) provided at least 8 hours of data on 3 weekdays and 1 weekend day.
Measure: Mean (Standard Deviation); unit: mean minutes per hour
Arm/Group | Control | Physical Activity Intervention
Number analyzed (Participants) | 680 | 706
mean minutes per hour | 3.27 (1.49) | 3.27 (1.49)
Statistical Analysis 1: Comparison: Control vs Physical Activity Intervention; Hypotheses: Post-intervention, weighted mean minutes of MVPA/week will be greater by 16 minutes among girls in intervention than control schools. Mean minutes per week is determined by multiplying mean minutes/hour by 90 hours that girls are awake in a week (10 hours awake on each weekend day; 14 hours awake on each weekday); Test type: Equivalence — Linear mixed-effect models were applied to examine the intervention effect on MVPA at post-intervention. Models included the group variable, cluster random effect of school, and the following fixed effects: age, BMI z-score, race, SES, ethnicity, pubertal stage, and study year. Baseline MVPA was included when evaluating the intervention effect at post-intervention; p = .207, Mixed Models Analysis; parameter estimate = -0.08, 95% CI 2-sided [-0.21 to 0.05]

2. Secondary Outcome: Cardiovascular Fitness (Aerobic Performance)
Description: Between group comparison measured by number of laps run in a progressive shuttle run test. CV fitness was assessed via estimation of maximal oxygen consumption.
Time Frame: Cardiovascular fitness after 17-week intervention (post-intervention)
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Control | Physical Activity Intervention
Number analyzed (Participants) | 680 | 706
ml/kg/min | 37.32 (5.28) | 37.51 (5.19)
Statistical Analysis 1: Comparison: Control vs Physical Activity Intervention; Immediately post-intervention, cardiovascular (CV) fitness will be higher among girls in the intervention than control schools; Test type: Equivalence — Linear mixed models were used to analyze intervention effect on CV fitness according to intention-to-treat, with school pairs treated as random effect and students nested within school and treatment condition. Models included main intervention predictor (control or intervention), incorporated cluster random effect, specified school pairs (random intercept), and controlled for baseline CV fitness, physical activity, race, socioeconomic status, ethnicity, pubertal stage, and study year cohort; p = .018, Mixed Models Analysis; parameter estimate = 0.20, 95% CI 2-sided [0.03 to 0.36], Standard Error of Mean 0.08

3. Secondary Outcome: Body Mass Index (BMI) Z-score
Description: To obtain BMI-z score, height and weight were assessed. Height was measured to nearest 0.1 cm using portable stadiometer.
  Weight was assessed to nearest 0.1 kg with foot-to-foot bioelectric impedance analysis scale. BMI was calculated and then converted into a percentile using age- and sex-specific reference values from the Centers for Disease Control and Prevention growth charts to determine BMI-z score.
Time Frame: Body mass index z-score at post-intervention (after 17-week intervention)
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Control | Physical Activity Intervention
Number analyzed (Participants) | 680 | 706
z-score | 1.01 (0.01) | 0.99 (0.01)
Statistical Analysis 1: Comparison: Control vs Physical Activity Intervention; Immediately post-intervention, BMI z-score will be significantly lower among girls in the intervention than control schools; Test type: Other — Linear mixed models were used to analyze intervention effect on BMI-z according to intention-to-treat, with school pairs treated as random effect and students nested within school and treatment condition. Models for BMI-z included main intervention predictor (control or intervention), incorporated cluster random effect, specified school pairs (random intercept), and controlled for baseline BMI-z, physical activity, race, socioeconomic status, ethnicity, pubertal stage, and study year cohort; p = .191, Mixed Models Analysis; parameter estimate = -0.02, 95% CI 2-sided [-0.05 to 0.01], Standard Error of Mean 0.01

4. Secondary Outcome: Percent Body Fat
Description: Percent body fat estimated via a foot-to-foot body weight scale with bioelectrical impedance analysis capabilities.
Time Frame: Percent body fat at post-intervention (immediately after 17-week intervention)
Measure: Mean (Standard Error); unit: percent body fat
Arm/Group | Control | Physical Activity Intervention
Number analyzed (Participants) | 680 | 706
percent body fat | 30.67 (0.14) | 30.30 (0.14)
Statistical Analysis 1: Comparison: Control vs Physical Activity Intervention; Immediately post-intervention, percent body fat will be significantly lower among girls in the intervention than control schools; Test type: Equivalence — Linear mixed models were used to analyze intervention effect on % body fat according to intention-to-treat, with school pairs treated as random effect and students nested within school and treatment condition. Models included main intervention predictor (control or intervention), incorporated cluster random effect, specified school pairs (random intercept), and controlled for baseline % body fat, age, physical activity, race, socioeconomic status, ethnicity, pubertal stage, and year cohort; p = .007, Mixed Models Analysis; parameter estimate = -0.37, 95% CI 2-sided [-0.64 to -0.10], Standard Error of Mean 0.14

5. Other Pre Specified Outcome: Minutes of Moderate-to-Vigorous Physical Activity 9-month Follow up
Description: Minutes of MVPA were measured via ActiGraph GT3X+ accelerometers worn on an elastic belt at the right hip for 7 consecutive days, including 5 weekdays and 2 weekend days at 9-month follow up. Monitors were set to start collecting and storing data in raw format beginning 5:00 A.M. on the day after they were distributed to girls each school. Data were re-integrated to 15-second epochs and processed using established intensity cut-points. One week after distribution, data collectors returned to each school to collect the accelerometers. An imputation approach based on all available data in hour blocks on all 7 days was implemented. Wear time was standardized to 14 hours/weekday (one hour before each school's actual start time; 7 hours during school; 6 hours after school) and 10 hours/weekend day (later awake time from 11 a.m. to 9 p.m.).
Time Frame: 9 months after the end of the 17-week intervention
Measure: Mean (Standard Deviation); unit: mean minutes per hour
Groups:
- Control: The control group received usual school activities and wore accelerometers 9-months after the Girls on the Move intervention had ended.
- Physical Activity Intervention: The intervention group wore accelerometers to measure MVPA 9 months after the Girls on the Move intervention had ended.
Arm/Group | Control | Physical Activity Intervention
Number analyzed (Participants) | 766 | 753
mean minutes per hour | 2.64 (1.15) | 2.59 (1.19)
Statistical Analysis 1: Comparison: Control vs Physical Activity Intervention; Test type: Equivalence — Linear mixed-effect models were applied to examine the intervention effect on MVPA at 9-month follow up. Models included the group variable, cluster random effect of school, and the following fixed effects: age, BMI z-score, race, SES, ethnicity, pubertal stage, and study year. Baseline MVPA was included when evaluating the intervention effect at follow up; p = .118, Mixed Models Analysis; parameter estimate = -0.09, 95% CI 2-sided [-0.21 to 0.02]

6. Other Pre Specified Outcome: Perceived Benefits of Physical Activity
Description: To assess positive consequences of physical activity, girls completed 10-item Perceived Benefits Scale. Response choices ranged form (0) not at all true to (3) very true. Higher score means better outcome.
Time Frame: baseline to post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control: Received usual school activities
- Intervention: Received Girls on the Move intervention
Arm/Group | Control | Intervention
Number analyzed (Participants) | 766 | 753
score on a scale | 2.22 (0.51) | 2.29 (0.53)
Statistical Analysis 1: Comparison: Control vs Intervention; Path analysis was performed to examine study mediation model. Maximum likelihood estimates were computed. Model fit was evaluated based on fit indices: (a) Goodness-of-Fit Index (GFI) ≥.95, (b) Comparative Fit Index (CFI) ≥.95, (c) Root Mean Square Error of Approximation (RMSEA) ≤.05; (d) standardized root mean squared residual (SRMR) ≤.08; and (e) chi-square test p>.05.26; Test type: Other; parameter estimate = -.97

7. Other Pre Specified Outcome: Perceived Barriers to Physical Activity
Description: To assess obstacles interfering with physical activity, girls completed a 16-item Perceived Barriers Scale. Response choices ranged from (0) not at all true to (3) very true. Higher score means worse outcome.
Time Frame: Baseline to post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control: Usual school activities
- Intervention: Received intervention
Arm/Group | Control | Intervention
Number analyzed (Participants) | 766 | 753
score on a scale | 1.14 (0.60) | 1.26 (0.63)
Statistical Analysis 1: Comparison: Control vs Intervention; Path analysis was performed to examine study mediation model. Maximum likelihood estimates were computed. Model fit was evaluated based on fit indices: (a) Goodness-of-Fit Index (GFI) ≥.95, (b) Comparative Fit Index (CFI) ≥.95, (c) Root Mean Square Error of Approximation (RMSEA) ≤.05; (d) standardized root mean squared residual (SRMR) ≤.08; and (e) chi-squar; Test type: Other; parameter estimate = 2.90

8. Other Pre Specified Outcome: Physical Activity Self-Efficacy
Description: To measure girls' confidence in their ability to attain physical activity during their free time when facing barriers or not, a 6-item Physical Activity Self-Efficacy scale was used. Response choices ranged from (0) disagree a lot to (3) agree a lot. Higher score means better outcome.
Time Frame: baseline to post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control: Usual activities
Arm/Group | Control | Intervention
Number analyzed (Participants) | 766 | 753
score on a scale | 2.14 (0.60) | 2.12 (0.64)
Statistical Analysis 1: Comparison: Control vs Intervention; [analysis description as in outcome 7, analysis 1]; Test type: Other; parameter estimate = .47

9. Other Pre Specified Outcome: Social Support for Physical Activity
Description: To measure assistance for physical activity received form others, an 8-item Social Support Scale was used. Response choices ranged form (0) never to (3) often. Higher score means better outcome.
Time Frame: baseline to post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 766 | 753
score on a scale | 1.73 (0.86) | 1.87 (0.82)
Statistical Analysis 1: Comparison: Control vs Intervention; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < .001, Path analysis; parameter estimate = 30.48

10. Other Pre Specified Outcome: Enjoyment of Physical Activity
Description: To assess feelings or fun regarding physical activity, a 6-item Physical Activity Enjoyment Scale was used. Response choices ranged form (0) not at all true to (3) very true. Higher score means better outcome.
Time Frame: baseline to post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 766 | 753
score on a scale | 2.11 (0.72) | 2.11 (0.67)
Statistical Analysis 1: Comparison: Control vs Intervention; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < .001, Path analysis; parameter estimate = 24.48

11. Other Pre Specified Outcome: Motivation for Physical Activity
Description: To assess feelings regarding physical activity, a 10-item scale was used. Response choices ranged from (0) not true to (4) very true. Higher score means better outcome.
Time Frame: baseline to post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 766 | 753
score on a scale | 3.48 (0.69) | 3.48 (0.68)
Statistical Analysis 1: Comparison: Control vs Intervention; [analysis description as in outcome 7, analysis 1]; Test type: Other; parameter estimate = 3.19

ADVERSE EVENTS:
Time Frame: From baseline data collection through post-intervention data collection after the 17-week intervention to 9-month post-intervention follow up (1 year, 2 months)
Arm/Group | Control | Physical Activity Intervention
Serious Adverse Events (participants affected / at risk) | 0/777 | 0/766
Other Adverse Events (participants affected / at risk) | 0/777 | 0/766

LIMITATIONS AND CAVEATS:
Costs were not analyzed. Attendance at the physical activity (PA) club was less than optimal. Study lacked a plan for girls to sustain PA in post-intervention period. Generalizability may be limited (sample selected from certain geographical area).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No